CLINICAL TRIAL: NCT05478057
Title: Supplementary Motor Area is a Potential Target for Speech Disturbance in Parkinson Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202102465A3A0
Record Dates: First submitted 2022-07-11; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease
Keywords: speech disturbance; transcranial magnetic stimulation
MeSH Terms: conditions — Parkinson Disease; Speech Disorders | interventions — Transcranial Magnetic Stimulation; Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PD patients with speech disturbance treated with 10 Hz rTMS (Experimental)
  Interventions: Device: "MAGSTIM" Repetitive transcranial magnetic stimulator (rTMS) system
- PD patients with speech disturbance treated with sham rTMS (Sham Comparator)
  Interventions: Device: "MAGSTIM" Repetitive transcranial magnetic stimulator (rTMS) system
- PD patients without speech disturbance treated with 10 Hz rTMS (Experimental)
  Interventions: Device: "MAGSTIM" Repetitive transcranial magnetic stimulator (rTMS) system
- PD patients without speech disturbance with sham rTMS (Sham Comparator)
  Interventions: Device: "MAGSTIM" Repetitive transcranial magnetic stimulator (rTMS) system

INTERVENTIONS:
Device: "MAGSTIM" Repetitive transcranial magnetic stimulator (rTMS) system — we plan to recruit 60 patients with Parkinson disease, comprising 30 patients with speech disturbance and 30 age- and sex-match patients without speech disturbance. Each group of patients will be randomly divided into sham stimulation or rTMS. A total of 10 rTMS sessions will be applied in 2 weeks. The effect of rTMS will be evaluated via the changes of speech performance and functional connectivity which was analyzed from resting-state functional magnetic resonance imaging.

SUMMARY:
Speech disturbance is common in patients with Parkinson disease. Pharmacotherapy improves motor symptoms but has inconsistent effects on speech disturbance in PD patients. Transcranial magnetic stimulation (TMS) is a safe and non-invasive tool used for brain stimulation. Repetitive transcranial magnetic stimulation (rTMS) has positive effects on motor function of PD. Yet, its effect on speech disturbance seems to be inconclusive. Previous rTMS studies mainly focused on the primary motor cortex for PD speech disturbance. Nevertheless, we think supplementary motor area (SMA) may be a better target. Speech disturbance in PD may be associated with basal ganglia-thalamocortical motor circuits and SMA involves in the cortex part. In addition, neuroimaging studies showed that SMA were under-activation in PD patients. Therefore, we conduct this 3-year study including two experiments. The aim of the study is to determine if rTMS over SMA can improve the speech function of PD patients and change the functional connectivity of speech pathway in the brain. This will be the first study to investigate the effect of rTMS over SMA on speech.

ELIGIBILITY:
Experiment 1

Inclusion Criteria:

* right-handed healthy adult volunteers who understand and agree on the informed consent of the study

Exclusion Criteria:

* pregnancy or possibility of pregnancy
* history of seizure
* family history of epilepsy
* metals in any part of the body.

Experiment 2

Inclusion Criteria:

* PD patients with speech disturbance who understand and agree on the informed consent of the study. The speech item scored 2 or 3 in the unified Parkinson's disease rating scale (UPDRS) part III.

Exclusion Criteria:

* dementia
* the history of stroke, brain lesion, other central nervous system diseases
* the contraindication of TMS which described above
* any contraindication of MRI

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of speech performance from baseline in experiment 1 | Baseline ((1) before rTMS), (2) immediately after rTMS
  1. sustained phonation of /a/ for as long and steady as possible in one breath
  2. fast pa-/ta-/ka- repetition at least nine times in one breath
  3. reading a standardized paragraph composed of 80 words as clear and fast as possible
Change of speech performance from baseline in experiment 2 | Baseline ((1) before rTMS), (2) within 24 hours after 10 times of rTMS (3) 8 weeks later after 10 times of rTMS
  1. sustained phonation of /a/ for as long and steady as possible in one breath
  2. fast pa-/ta-/ka- repetition at least nine times in one breath
  3. reading a standardized paragraph composed of 80 words as clear and fast as possible
Change of functional connectivity from baseline in experiment 2 | Baseline ((1) before rTMS), (2) within 24 hours after 10 times of rTMS
  use rs-fMRI to compare the functional connectivity between PD patients with and without speech disturbance and the changes of connectivity after rTMS over SMA